CLINICAL TRIAL: NCT03437434
Title: Gore-Tex Suture and BunnyLens Scleral Fixation - Historical Retrospective Trial
Brief Title: Scleral Fixation of BunnyLens With GoreTex Suture- Initial Results
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DAVID HAUSER (Other)
Responsible Party: Sponsor-Investigator, DAVID HAUSER, Retina Ophthalmologist, Barzilai Medical Center
Organization: Barzilai Medical Center (Other)
Other Study IDs: 114-16-BRZ
Record Dates: First submitted 2018-01-21; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Aphakia, Acquired
MeSH Terms: conditions — Aphakia | interventions — Visual Acuity; Refraction, Ocular; Microscopy, Acoustic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BunnyLens and Gore-Tex suture: All patients Underwent 4 point PC-IOL scleral fixation with Gore-Tex sutures
  Interventions: Other: Visual Acuity

INTERVENTIONS:
Other: Visual Acuity — Ocular Examination
  Other Names: Refraction; Biomicroscopy

SUMMARY:
This study evaluates the Visual Acuity and refraction of patients post 4-point Scleral fixation of BunnyLens (Intra Ocular Lens- IOL) with GoreTex sutures. All patients underwent secondary IOL implantation or IOL exchange during 2014-2017.

DETAILED DESCRIPTION:
4 point scleral fixation of PC- IOL (Posterior Chamber-PC) BunnyLens with Gore-Tex sutures is a surgical technique for implanting IOL in patients with capsular support absence, due to trauma, abnormal anterior chamber, IOL dislocation, or ciliary zonule defect.

The 4 point fixation enables to align the PC- IOL with minimal vertical and horizontal deviation;The Gore-Tex sutures maintain stable scleral fixation with no suture erosion or breakage.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent secondary cataract surgery or IOL replacement and BunnyLens fixation with Gore-Tex sutures.

Exclusion Criteria:

* Lack of Cooperation, death, severe physical or mental illness, patient's request to withdraw of the clinical trial.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are capable of inform consent and are eligible according to the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-03-24 (Estimated); Study Completion 2018-04-24 (Estimated)

PRIMARY OUTCOMES:
Distance Visual Acuity | Up to 24 months from surgery.
  Degree of Visual Acuity is measured in LogMar (-0.3 to1) and by Decimal Value (0.0-2.0)
Ocular Refraction | Up to 24 months from surgery.
  Refraction of the Ocular surfaces, measured in sphere, cylinder and axis.

SECONDARY OUTCOMES:
Slit Lamp Biomicroscopy | Up to 24 months from surgery.
  Slit lamp examination of the anterior and posterior segments.

CONTACTS AND LOCATIONS:
Overall Officials: David Hauser, MD, Principal Investigator — Barzilai University Medical Center
Locations (1):
- Barzilai University Medical Center, Ashkelon, Israel